CLINICAL TRIAL: NCT04548063
Title: Consent Forms in Cancer Research: Examining the Effect of Length on Readability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20-007236
Record Dates: First submitted 2020-09-09; First posted 2020-09-14 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6,000 word consent form (Experimental): Subjects who are receiving cancer therapy or have been treated for cancer in the past will be asked to review a mock consent form of approximately 6,000 words.
  Interventions: Other: 6,000 word consent form
- 4,000 word consent form (Experimental): Subjects who are receiving cancer therapy or have been treated for cancer in the past will be asked to review a mock consent form of approximately 4,000 words.
  Interventions: Other: 4,000 word consent form
- 2,000 word consent form (Experimental): Subjects who are receiving cancer therapy or have been treated for cancer in the past will be asked to review a mock consent form of approximately 2,000 words.
  Interventions: Other: 2,000 word consent form

INTERVENTIONS:
Other: 6,000 word consent form — Mock consent form with consistent content in approximately 6,000 word length.
  Arms: 6,000 word consent form
Other: 4,000 word consent form — Mock consent form with consistent content in approximately 4,000 word length.
  Arms: 4,000 word consent form
Other: 2,000 word consent form — Mock consent form with consistent content in approximately 2,000 word length.
  Arms: 2,000 word consent form

SUMMARY:
Researchers are using mock consent forms to see if wordiness has any effect on patients' understanding and willingness to sign up for a cancer clinical trial.

DETAILED DESCRIPTION:
This study will determine whether there is a relationship between wordiness of a consent form and whether or not the consent form helped the patient decide to enroll in a clinical trial. This study will also determine whether wordiness of a consent form is associated with patients' willingness to sign the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patient-reported history of cancer
* Patient is able to read English
* Patient-reported age of 18 years or older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Decision to enroll | Through study completion, approximately 1 hour
  Number of participants to indicate on the self-reported patient questionnaire that the information provided in the consent form helped make a decision about whether or not to enroll in the trial. This is defined as a response of 1 or 2 on the Likert scale of 1=strongly agree and 5= strongly disagree for information in the consent form was helpful to the decision to join the study.

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almodallal Y, Duong Q, Satele D, Novotny P, Cook KD, Chauhan C, Daiss MK, Le-Rademacher J, Looker S, Martin N, Smestad MF, Winham SJ, Mandrekar SJ, Jatoi A. Randomized, Double-Blind Trial on the Impact of Word Count in Cancer Clinical Trial Consent Forms. JCO Oncol Pract. 2021 Oct;17(10):e1460-e1472. doi: 10.1200/OP.21.00071. Epub 2021 Jun 14. PMID 34125586
- [Background] Wieland J, Satele D, Almodallal Y, Novotny P, Pritzl SL, Mandrekar SJ, Jatoi A. Succinct Cancer Clinical Trial Consent Forms in Rural Patients With Cancer: A Secondary Analysis of a Randomized, Double-Blinded study. J Patient Exp. 2022 Jun 22;9:23743735221107242. doi: 10.1177/23743735221107242. eCollection 2022. PMID 35756962
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials